CLINICAL TRIAL: NCT02935634
Title: A Phase 2, Fast Real-time Assessment of Combination Therapies in Immuno-ONcology Study in Participants With Advanced Gastric Cancer (FRACTION-Gastric Cancer)
Brief Title: A Study to Test Combination Treatments in Participants With Advanced Gastric Cancer
Acronym: FRACTION-GC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA018-003; 2016-002807-24 (EudraCT Number)
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab; relatlimab; linrodostat; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Nivolumab + Ipilimumab (Active Comparator)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab + Relatlimab (Experimental)
  Interventions: Biological: Nivolumab; Biological: Relatlimab
- Nivolumab + BMS-986205 (Experimental)
  Interventions: Biological: Nivolumab; Biological: BMS-986205
- Nivolumab + Rucaparib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Rucaparib
- Ipilimumab + Rucaparib (Experimental)
  Interventions: Biological: Ipilimumab; Drug: Rucaparib
- Nivolumab + Ipilimumab + Rucaparib (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Drug: Rucaparib

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Nivolumab + BMS-986205; Nivolumab + Ipilimumab; Nivolumab + Ipilimumab + Rucaparib; Nivolumab + Relatlimab; Nivolumab + Rucaparib
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Ipilimumab + Rucaparib; Nivolumab + Ipilimumab; Nivolumab + Ipilimumab + Rucaparib
Biological: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016
  Arms: Nivolumab + Relatlimab
Biological: BMS-986205 — Specified dose on specified days
  Arms: Nivolumab + BMS-986205
Drug: Rucaparib — Specified dose on specified days
  Other Names: Rubraca
  Arms: Ipilimumab + Rucaparib; Nivolumab + Ipilimumab + Rucaparib; Nivolumab + Rucaparib

SUMMARY:
The purpose of this study is to evaluate the preliminary efficacy, safety, and tolerability of Nivolumab in combination with Ipilimumab or other treatment therapies in participants with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable, advanced or metastatic esophageal cancer (EC), gastric cancer (GC) or gastroesophageal junction (GEJ) carcinoma and have histologically confirmed predominant adenocarcinoma and/or squamous carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* At least 1 lesion with measurable disease

Exclusion Criteria:

* HER2-positive tumor and previously untreated with trastuzumab
* Suspected, known or progressive central nervous system metastases
* Other active malignancy requiring concurrent intervention
* Active, known or suspected autoimmune disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (16):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Local Institution - 0020, Duarte, California
  - University Of Colorado, Aurora, Colorado
  - Local Institution - 0032, New Haven, Connecticut
  - Local Institution - 0036, Washington D.C., District of Columbia
  - UF Health Medical Oncology - Davis Cancer Pavilion, Gainesville, Florida
  - Local Institution - 0038, Jacksonville, Florida
  - Local Institution - 0006, Baltimore, Maryland
  - Local Institution - 0017, Rochester, Minnesota
  - Local Institution - 0003, St Louis, Missouri
  - Local Institution - 0001, Hackensack, New Jersey
  - Local Institution - 0007, New York, New York
  - Local Institution - 0002, Portland, Oregon
  - Local Institution - 0005, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Local Institution - 0004, Seattle, Washington
- Australia (3):
  - Local Institution - 0035, Westmead, New South Wales
  - Local Institution - 0033, Heidelberg, Victoria
  - Local Institution, Randwick
- Canada (5):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Ottawa, Ontario
  - Local Institution - 0025, Toronto, Ontario
  - Local Institution - 0021, Toronto, Ontario
- Germany (2):
  - Local Institution - 0039, Heidelberg
  - Local Institution - 0043, Leipzig
- Israel (2):
  - Local Institution, Ramat Gan
  - Local Institution, Tel Aviv
- Italy (2):
  - Local Institution - 0014, Milan, Lombardy
  - IRCCS Istituto Nazionale Tumori Milano, Milan
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Utrecht
- Local Institution - 0050, Singapore, Singapore
- Switzerland (2):
  - Local Institution - 0041, Chur, Graubünden (de)
  - Local Institution - 0042, Zurich

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 190 participants that were randomized, 104 were initially randomized to Track 1 and 86 were initially randomized to Track 2. The 93 participants that started treatment in Track 2 include the total number of participants that received treatment in each arm which incorporates the 20 participants from Track 1 or 2 that were re-randomized to receive a different treatment combination in Track 2.
Groups:
- Nivolumab + Ipilimumab: Participants received nivolumab 1 mg/kg via IV infusion followed by ipilimumab 3 mg/kg administered IV Q3W, followed 6 weeks after the last dose of combination study treatment by nivolumab 480 mg administered IV Q4W for 2 years.
- Nivolumab + BMS-986016: Participants received nivolumab 240 mg via IV infusion Q2W followed by BMS-986016 80 mg administered IV Q2W for 2 years.
- Nivolumab + BMS-986205: Participants received nivolumab 480 mg Q4W and BMS-986205 100 mg QD for 104 weeks.
- Nivolumab + Rucaparib: Participants received nivolumab 480 mg administered IV Q4W in combination with rucaparib 600 mg administered orally twice daily for 2 years.
- Ipilimumab + Rucaparib: Participants received ipilimumab 3 mg/kg administered IV Q4W in combination with rucaparib 600 mg orally twice daily for 2 years.
- Nivolumab + Ipilimumab + Rucaparib: Participants received nivolumab 480 mg administered IV Q4W in combination with ipilimumab 1 mg/kg administered IV Q6W and rucaparib 600 mg orally twice daily for 2 years.
Period: Randomization
Arm/Group | Nivolumab + Ipilimumab | Nivolumab + BMS-986016 | Nivolumab + BMS-986205 | Nivolumab + Rucaparib | Ipilimumab + Rucaparib | Nivolumab + Ipilimumab + Rucaparib
Started | 42 | 54 | 62 | 12 | 10 | 10
Randomized to Track 1 | 23 | 22 | 38 | 7 | 8 | 6
Randomized to Track 2 | 19 | 32 | 24 | 5 | 2 | 4
Completed | 40 | 50 | 59 | 12 | 10 | 10
Not Completed | 2 | 4 | 3 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Other reasons | 0 | 2 | 2 | 0 | 0 | 0
Period: Treatment: Track 1
Arm/Group | Nivolumab + Ipilimumab | Nivolumab + BMS-986016 | Nivolumab + BMS-986205 | Nivolumab + Rucaparib | Ipilimumab + Rucaparib | Nivolumab + Ipilimumab + Rucaparib
Started (Treatment naive participants) | 23 | 20 | 38 | 7 | 8 | 6
Re-Randomized to Track 2 | 2 | 3 | 3 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 0 | 0 | 0
Not Completed | 22 | 19 | 37 | 7 | 8 | 6
Not completed — Disease progression | 15 | 17 | 28 | 4 | 6 | 2
Not completed — Adverse event unrelated to study drug | 1 | 1 | 2 | 3 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study drug toxicity | 2 | 1 | 3 | 0 | 0 | 1
Not completed — Participant request to discontinue treatment | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Participant withdrew consent | 2 | 0 | 1 | 0 | 1 | 0
Not completed — Other reasons | 0 | 0 | 2 | 0 | 0 | 0
Period: Treatment: Track 2
Arm/Group | Nivolumab + Ipilimumab | Nivolumab + BMS-986016 | Nivolumab + BMS-986205 | Nivolumab + Rucaparib | Ipilimumab + Rucaparib | Nivolumab + Ipilimumab + Rucaparib
Started (Treatment experienced participants) | 23 | 36 | 22 | 6 | 2 | 4
No Pre-Randomization | 17 | 30 | 21 | 5 | 2 | 4
Re-Randomized From Track 1 Nivolumab + Relatlimab | 1 | 0 | 1 | 1 | 0 | 0
Re-Randomized From Track 1 Nivolumab + Ipilimumab | 2 | 1 | 0 | 0 | 0 | 0
Re-Randomized From Track 2 Nivolumab + Relatlimab | 0 | 2 | 0 | 0 | 0 | 0
Re-Randomized From Track 2 Nivolumab + BMS986205 | 3 | 0 | 0 | 0 | 0 | 0
Previously Un-Treated But Re-Randomized | 0 | 1 | 0 | 0 | 0 | 0
Re-Randomized From Track 2 Nivolumab + Ipilimumab | 0 | 2 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 0 | 1 | 0 | 0
Not Completed | 22 | 34 | 22 | 5 | 2 | 4
Not completed — Disease progression | 13 | 26 | 20 | 5 | 1 | 4
Not completed — Adverse event unrelated to study drug | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Study drug toxicity | 7 | 3 | 0 | 0 | 0 | 0
Not completed — Participant request to discontinue treatment | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Track 1: Nivolumab + Ipilimumab: Treatment naive participants received nivolumab 1 mg/kg via IV infusion followed by ipilimumab 3 mg/kg administered IV Q3W, followed 6 weeks after the last dose of combination study treatment by nivolumab 480 mg administered IV Q4W for 2 years.
- Track 1: Nivolumab + BMS-986016: Treatment naive participants received nivolumab 240 mg via IV infusion Q2W followed by BMS-986016 80 mg administered IV Q2W for 2 years.
- Track 1: Nivolumab + BMS-986205: Treatment naive participants received nivolumab 480 mg Q4W and BMS-986205 100 mg QD for 104 weeks.
- Track 1: Nivolumab + Rucaparib: Treatment naive participants received nivolumab 480 mg administered IV Q4W in combination with rucaparib 600 mg administered orally twice daily for 2 years.
- Track 1: Ipilimumab + Rucaparib: Treatment naive participants received ipilimumab 3 mg/kg administered IV Q4W in combination with rucaparib 600 mg orally twice daily for 2 years.
- Track 1: Nivolumab + Ipilimumab + Rucaparib: Treatment naive participants received nivolumab 480 mg administered IV Q4W in combination with ipilimumab 1 mg/kg administered IV Q6W and rucaparib 600 mg orally twice daily for 2 years.
- Track 2: Nivolumab + Ipilimumab: Treatment experienced participants received nivolumab 1 mg/kg via IV infusion followed by ipilimumab 3 mg/kg administered IV Q3W, followed 6 weeks after the last dose of combination study treatment by nivolumab 480 mg administered IV Q4W for 2 years.
- Track 2: Nivolumab + BMS-986016: Treatment experienced participants received nivolumab 240 mg via IV infusion Q2W followed by BMS-986016 80 mg administered IV Q2W for 2 years.
- Track 2: Nivolumab + BMS-986205: Treatment experienced participants received nivolumab 480 mg Q4W and BMS-986205 100 mg QD for 104 weeks.
- Track 2: Nivolumab + Rucaparib: Treatment experienced participants received nivolumab 480 mg administered IV Q4W in combination with rucaparib 600 mg administered orally twice daily for 2 years.
- Track 2: Ipilimumab + Rucaparib: Treatment experienced participants received ipilimumab 3 mg/kg administered IV Q4W in combination with rucaparib 600 mg orally twice daily for 2 years.
- Track 2: Nivolumab + Ipilimumab + Rucaparib: Treatment experienced participants received nivolumab 480 mg administered IV Q4W in combination with ipilimumab 1 mg/kg administered IV Q6W and rucaparib 600 mg orally twice daily for 2 years.
- Total: Total of all reporting groups
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib | Total
Number analyzed (Participants) | 23 | 22 | 38 | 7 | 8 | 6 | 19 | 32 | 24 | 5 | 2 | 4 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (11.0) | 58.1 (12.6) | 60.6 (12.9) | 58.1 (10.4) | 57.4 (13.9) | 59.5 (6.7) | 55.9 (12.0) | 61.8 (11.8) | 64.2 (9.2) | 58.0 (16.2) | 57.0 (2.8) | 53.0 (16.4) | 60.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 14 | 0 | 4 | 2 | 2 | 7 | 9 | 1 | 0 | 0 | 48
  Male | 18 | 18 | 24 | 7 | 4 | 4 | 17 | 25 | 15 | 4 | 2 | 4 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 13 | 17 | 17 | 2 | 2 | 4 | 14 | 25 | 17 | 3 | 2 | 2 | 118
  Unknown or Not Reported | 9 | 5 | 20 | 5 | 6 | 2 | 4 | 7 | 6 | 2 | 0 | 2 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 22 | 19 | 32 | 7 | 7 | 6 | 13 | 29 | 19 | 4 | 1 | 3 | 162
    Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 9
    Asian | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 9
    American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Other | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 6
    Not reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Investigator
Description: ORR is the percent of participants whose best overall response (BOR) is complete response (CR) or partial response (PR). BOR is the best response from the start of the study treatment until objectively documented progression per RECIST v1.1 or subsequent anticancer therapy, whichever occurs first. CR is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The Response Evaluation Criteria in Solid Tumors (RECIST) is a standard way to measure the response of a tumor to treatment. CR+PR, confidence interval based on Clopper and Pearson method.
Time Frame: From first dose of study treatment until progression or subsequent anticancer therapy, whichever occurs first (up to approximately 65 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib
Number analyzed (Participants) | 23 | 20 | 38 | 7 | 8 | 6 | 23 | 36 | 22 | 6 | 2 | 4
Percent of participants | 4.3 [0.1 to 21.9] | 5.0 [0.1 to 24.9] | 13.2 [4.4 to 28.1] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9] | 16.7 [0.4 to 64.1] | 8.7 [1.1 to 28.0] | 5.6 [0.7 to 18.7] | 0 [0.0 to 15.4] | 0 [0.0 to 45.9] | 0 [0.0 to 84.2] | 0 [0.0 to 60.2]

2. Primary Outcome: Median Duration of Response (DOR)
Description: Duration of Response (DOR) is the time between the date of first response and the date of first documented disease progression as determined by RECIST 1.1 or death due to any cause, whichever occurred first. Complete Response (CR) is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Median computed using Kaplan -Meier method.
Time Frame: From first dose to date of first documented tumor progression or death due to any cause, whichever occurred first (up to approximately 65 months)
Population: All treated participants with a complete response (CR) or partial response (PR)
Measure: Median (Full Range); unit: Weeks
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib
Number analyzed (Participants) | 1 | 1 | 5 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Weeks | 156.0 [156.0 to 156.0] | NA [113.4 to 113.4] — Unable to calculate DOR due to insufficient number of participants who responded | NA [37.3 to 144.0] — Unable to calculate DOR due to insufficient number of participants who responded |  |  | NA [0.1 to 0.1] — Unable to calculate DOR due to insufficient number of participants who responded | 14.71 [0.1 to 14.71] | 16.86 [8.1 to 25.6] |  |  |  |

3. Primary Outcome: Kaplan-Meier Analysis of Progression Free Survival Rate (PFSR) at 24 Weeks
Description: The PFSR at 24 weeks is defined as the proportion of treated participants remaining progression free and surviving at 24 weeks since the first dosing date. Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Point estimates are derived from Kaplan-Meier analyses, the 95% CIs are derived from Greenwood formula.
Time Frame: 24 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib
Number analyzed (Participants) | 23 | 20 | 38 | 7 | 8 | 6 | 23 | 36 | 22 | 6 | 2 | 4
Proportion of participants | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 0.240 [0.114 to 0.393] | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 0.170 [0.063 to 0.322] | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

4. Secondary Outcome: Number of Participants With AEs, SAEs, AEs Leading to Discontinuation, and Death
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose to 100 days after last dose of study therapy (assessed up to approximately 30 months)
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib
Number analyzed (Participants) | 23 | 20 | 38 | 7 | 8 | 6 | 23 | 36 | 22 | 6 | 2 | 4
Participants
  Adverse Events (AEs) | 23 | 20 | 38 | 7 | 8 | 6 | 23 | 36 | 22 | 6 | 2 | 4
  Serious Adverse Events (SAEs) | 19 | 15 | 24 | 5 | 6 | 4 | 17 | 24 | 12 | 4 | 2 | 3
  AEs Leading to Discontinuation | 9 | 7 | 11 | 3 | 4 | 4 | 10 | 8 | 2 | 0 | 1 | 0
  Death | 19 | 15 | 26 | 7 | 5 | 4 | 19 | 26 | 13 | 3 | 2 | 3

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: The number of participants with laboratory abnormalities in specific thyroid tests based on US conventional units. TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal.
Time Frame: From first dose to 100 days after last dose of study therapy (approximately 30 months)
Population: All treated participants with at least one on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib
Number analyzed (Participants) | 18 | 16 | 26 | 6 | 3 | 3 | 22 | 27 | 18 | 5 | 1 | 3
Participants
  TSH > ULN | 4 | 4 | 6 | 1 | 1 | 1 | 11 | 5 | 5 | 0 | 1 | 1
  TSH > ULN WITH TSH <= ULN AT BASELINE | 3 | 3 | 4 | 0 | 1 | 1 | 6 | 1 | 4 | 0 | 1 | 0
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 1 | 2 | 2 | 0 | 1 | 1 | 5 | 2 | 2 | 0 | 0 | 1
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 1 | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 2 | 1 | 3 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 1 | 0
  TSH < LLN | 1 | 2 | 5 | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0
  TSH <LLN WITH TSH >= LLN AT BASELINE | 0 | 1 | 3 | 0 | 0 | 0 | 3 | 5 | 0 | 0 | 0 | 0
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: The number of participants with laboratory abnormalities in specific liver tests based on US conventional units. ALT = Alanine Aminotransferase AST = Aspartate Aminotransferase ULN = Upper Limit of Normal
Time Frame: From first dose to 100 days after last dose of study therapy (approximately 30 months)
Population: All treated participants with at least one on-treatment AST, ALT and/or bilirubin test measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib
Number analyzed (Participants) | 19 | 20 | 33 | 6 | 8 | 4 | 22 | 32 | 22 | 6 | 2 | 3
Participants
  ALT OR AST > 3XULN | 6 | 6 | 5 | 1 | 2 | 1 | 6 | 2 | 2 | 3 | 1 | 0
  ALT OR AST> 5XULN | 3 | 2 | 3 | 0 | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 0
  ALT OR AST> 10XULN | 2 | 1 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
  ALT OR AST > 20XULN | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 19 | 20 | 33 | 6 | 7 | 4 | 22 | 32 | 22 | 6 | 2 | 3
  TOTAL BILIRUBIN > 2XULN | 2 | 3 | 0 | 1 | 1 | 1 | 3 | 1 | 3 | 1 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY: number analyzed (Participants) | 19 | 20 | 33 | 6 | 7 | 4 | 22 | 32 | 22 | 6 | 2 | 3
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 2 | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS: number analyzed (Participants) | 19 | 20 | 33 | 6 | 7 | 4 | 22 | 32 | 22 | 6 | 2 | 3
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 2 | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization until their study completion (up to approximately 65 months). SAEs and other AEs were assessed from first dose to 100 days after last dose of study therapy (up to approximately 30 months).
Description: The total number at risk for all-cause mortality represents all participants who were randomized and re-randomized. The total number at risk by any serious adverse event and other (not including serious) adverse events represents all participants who received at least 1 dose of study medication.
Arm/Group | Track 1: Nivolumab + Ipilimumab | Track 1: Nivolumab + BMS-986016 | Track 1: Nivolumab + BMS-986205 | Track 1: Nivolumab + Rucaparib | Track 1: Ipilimumab + Rucaparib | Track 1: Nivolumab + Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab | Track 2: Nivolumab + BMS-986016 | Track 2: Nivolumab + BMS-986205 | Track 2: Nivolumab + Rucaparib | Track 2: Ipilimumab + Rucaparib | Track 2: Nivolumab + Ipilimumab + Rucaparib
All-Cause Mortality (participants affected / at risk) | 19/23 | 15/23 | 26/39 | 7/7 | 5/8 | 4/6 | 19/28 | 26/41 | 13/25 | 3/6 | 2/2 | 3/4
Serious Adverse Events (participants affected / at risk) | 19/23 | 15/20 | 24/38 | 5/7 | 6/8 | 4/6 | 17/23 | 24/36 | 12/22 | 4/6 | 2/2 | 3/4
Other Adverse Events (participants affected / at risk) | 21/23 | 20/20 | 38/38 | 7/7 | 8/8 | 6/6 | 23/23 | 34/36 | 21/22 | 6/6 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Track 1: Nivolumab + Ipilimumab (N=23) | Track 1: Nivolumab + BMS-986016 (N=20) | Track 1: Nivolumab + BMS-986205 (N=38) | Track 1: Nivolumab + Rucaparib (N=7) | Track 1: Ipilimumab + Rucaparib (N=8) | Track 1: Nivolumab + Ipilimumab + Rucaparib (N=6) | Track 2: Nivolumab + Ipilimumab (N=23) | Track 2: Nivolumab + BMS-986016 (N=36) | Track 2: Nivolumab + BMS-986205 (N=22) | Track 2: Nivolumab + Rucaparib (N=6) | Track 2: Ipilimumab + Rucaparib (N=2) | Track 2: Nivolumab + Ipilimumab + Rucaparib (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 4 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 6 | 11 | 0 | 3 | 0 | 5 | 9 | 8 | 2 | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Superior vena cava stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Track 1: Nivolumab + Ipilimumab (N=23) | Track 1: Nivolumab + BMS-986016 (N=20) | Track 1: Nivolumab + BMS-986205 (N=38) | Track 1: Nivolumab + Rucaparib (N=7) | Track 1: Ipilimumab + Rucaparib (N=8) | Track 1: Nivolumab + Ipilimumab + Rucaparib (N=6) | Track 2: Nivolumab + Ipilimumab (N=23) | Track 2: Nivolumab + BMS-986016 (N=36) | Track 2: Nivolumab + BMS-986205 (N=22) | Track 2: Nivolumab + Rucaparib (N=6) | Track 2: Ipilimumab + Rucaparib (N=2) | Track 2: Nivolumab + Ipilimumab + Rucaparib (N=4)
Anaemia (Blood and lymphatic system disorders) | 6 | 8 | 12 | 1 | 3 | 2 | 7 | 11 | 7 | 1 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 3 | 4 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 7 | 11 | 2 | 1 | 2 | 7 | 6 | 1 | 3 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 2 | 0 | 0 | 2 | 1 | 2 | 3 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 5 | 9 | 2 | 2 | 2 | 7 | 6 | 4 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 7 | 4 | 1 | 2 | 7 | 7 | 3 | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 6 | 3 | 8 | 3 | 0 | 2 | 4 | 5 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jejunal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 10 | 17 | 4 | 4 | 2 | 10 | 9 | 6 | 4 | 0 | 2
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 5 | 7 | 0 | 1 | 2 | 7 | 7 | 1 | 2 | 0 | 2
Asthenia (General disorders) | 4 | 3 | 4 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Early satiety (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 13 | 11 | 23 | 2 | 5 | 2 | 10 | 22 | 11 | 5 | 2 | 2
General physical health deterioration (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 1 | 3 | 1 | 1 | 1 | 1 | 5 | 4 | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 7 | 3 | 8 | 1 | 2 | 0 | 4 | 5 | 2 | 2 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 5 | 7 | 1 | 3 | 4 | 5 | 3 | 2 | 1 | 1 | 0
Amylase increased (Investigations) | 1 | 3 | 4 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 8 | 2 | 3 | 4 | 5 | 3 | 4 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 5 | 3 | 1 | 2 | 6 | 4 | 4 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 6 | 3 | 2 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 3 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Lipase increased (Investigations) | 2 | 3 | 3 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 6 | 3 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 1 | 0
Weight decreased (Investigations) | 4 | 2 | 4 | 2 | 2 | 0 | 2 | 2 | 2 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 4 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 10 | 9 | 2 | 2 | 0 | 7 | 14 | 8 | 2 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 2 | 3 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 0 | 0 | 0 | 1 | 7 | 4 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 4 | 1 | 0 | 0 | 3 | 5 | 3 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 5 | 4 | 0 | 0 | 0 | 3 | 4 | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 0 | 0 | 1 | 5 | 3 | 2 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3 | 1 | 1 | 0 | 3 | 3 | 3 | 3 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 5 | 1 | 0 | 0 | 5 | 9 | 4 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 6 | 0 | 0 | 2 | 1 | 5 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 3 | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 8 | 1 | 0 | 1 | 4 | 7 | 3 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 7 | 0 | 1 | 0 | 5 | 6 | 1 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 5 | 1 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 0 | 1 | 2 | 6 | 4 | 2 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 0 | 3 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT02935634/Prot_SAP_000.pdf